CLINICAL TRIAL: NCT07274163
Title: Ambispective Registry of Patients Affected by Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Francesco Agustoni, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Lung Cancer Registry
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is one of the most common cancers and the leading cause of cancer-related death. It is often diagnosed late, and there are different types of lung cancer. Today, many patients benefit from targeted therapies and immunotherapy, which have improved survival.

This study will create an ambispective clinical registry of all lung cancer patients treated at Policlinico San Matteo.

The registry will collect data from 2019 to 2035 to better understand: 10-year overall survival, how the disease progresses over time, how patients respond to treatments and possible side effects, how patient and tumor characteristics influence treatment choices, how different therapies work in real-world practice.

All data will be securely collected whithin REDCap platform and used to improve future care and research.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years diagnosed with and/or treated for lung cancer at the department of SC Oncologia 1 Unit of the Fondazione IRCCS Policlinico San Matteo;
* Prospective patients (or their or legal guardians) who have the ability to understand and be willing to sign a written informed consent document;
* Retrospective patients who have signed the institutional document allowing the use of their data for research on their disease.

Exclusion Criteria:

* Patients who are unable to understand informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
10 years overall survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy